CLINICAL TRIAL: NCT02513121
Title: Randomized, Controlled Dietary Treatment Study of Pediatric NAFLD
Brief Title: Dietary Treatment Study of Pediatric NAFLD
Acronym: DTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Emory University (Other); Nutrition Science Initiative (Other)
Responsible Party: Principal Investigator, Jeffrey B. Schwimmer, MD, Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4405
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: NAFLD; Steatohepatitis; Nonalcoholic Steatohepatitis (NASH); Liver; Diet; Pediatric; Adolescent
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary modification (Active Comparator): Low free sugar diet
  Interventions: Other: Dietary modification
- Observational Arm (No Intervention): Standard of care

INTERVENTIONS:
Other: Dietary modification — The intervention is a modification of the family's habitual diet with a low sugar version of their diet.
  Arms: Dietary modification

SUMMARY:
This is an investigator initiated study being conducted in equal numbers at two sites, University of California, San Diego (UC San Diego) and Emory University (EU). The purpose of this study is to understand the potential of a low sugar diet for the treatment of nonalcoholic fatty liver disease (NAFLD) in children. Forty boys with NAFLD will be randomly assigned to either an intervention group or a habitual diet control group. The intervention will be a low sugar diet for a period of 8 weeks. The effect of this dietary change will be assessed using advanced magnetic resonance imaging (MRI) testing to measure liver fat.

ELIGIBILITY:
Inclusion Criteria:

* Boys age 11-16 years inclusive.
* Clinical history consistent with NAFLD.
* Biopsy-proven NAFLD
* MRI measured Liver Proton Density Fat Fraction ≥10%
* alanine aminotransferase (ALT) ≥ 45 u/L
* No evidence of any other liver disease by clinical history or histological evaluation.
* Written informed consent from parent or legal guardian.
* Written informed assent from the child or adolescent.

Exclusion Criteria:

Exclusions will not be based upon gender, race, or ethnicity. Participants with a current history of the following conditions or any other health issues that make it unsafe for them to participate in the opinion of the Investigators will be excluded from the study:

* History of significant alcohol intake (Alcohol Use Disorders Identification Test [AUDIT]) or inability to quantify alcohol consumption
* Chronic use (more than 2 consecutive weeks) of medications known to cause hepatic steatosis or steatohepatitis in the past year.
* The use of other known hepatotoxins within 120 days of baseline
* History of total parenteral nutrition (TPN) use in the year prior to screening
* History of bariatric surgery or planning to undergo bariatric surgery during the study duration
* Significant depression
* Non-compensated liver disease with any one of the following hematologic, biochemical, and serological criteria on entry into protocol:
* Hemoglobin < 10 g/dL
* White blood cell < 3,500 cells/mm
* Neutrophil count < 1,500 cells/mm3 of blood
* Platelets < 130,000 cells/mm3 of blood
* Direct bilirubin > 1.0 mg/dL
* Total bilirubin > 3 mg/dL
* Albumin < 3.2 g/dL
* International normalized ratio (INR) > 1.4
* Evidence of other chronic liver disease
* Children who are currently enrolled in a clinical trial or who received an investigational study drug or a medication with the intent to treat NAFLD/NASH in the past 60 days
* Contraindications to MRI, e.g. metal in the eyes, implanted electronic devices, aneurysm clips, pacemaker, cochlear implants
* Unable to have or complete the MRI exam due to body weight exceeding scanner table limit or girth exceeding scanner bore diameter
* Subjects who are not able or willing to comply with the protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator
* Families with > 5 individuals
* Failure to give informed consent

Ages: 11 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Schwimmer, MD, Principal Investigator — University of California, San Diego; Miriam Vos, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available in response to bona fide and good faith, ad hoc requests. Suitability of each request, if consistent with Institutional Review Board (IRB) approval, will be determined only in the case of a favorable vote of a majority of a committee consisting of each consortium investigator and the Grantor. Data will be made available with a signed access agreement.

REFERENCES:
- [Background] Schwimmer JB, Deutsch R, Rauch JB, Behling C, Newbury R, Lavine JE. Obesity, insulin resistance, and other clinicopathological correlates of pediatric nonalcoholic fatty liver disease. J Pediatr. 2003 Oct;143(4):500-5. doi: 10.1067/S0022-3476(03)00325-1. PMID 14571229
- [Background] Schwimmer JB, Deutsch R, Kahen T, Lavine JE, Stanley C, Behling C. Prevalence of fatty liver in children and adolescents. Pediatrics. 2006 Oct;118(4):1388-93. doi: 10.1542/peds.2006-1212. PMID 17015527
- [Background] Schwimmer JB, Pardee PE, Lavine JE, Blumkin AK, Cook S. Cardiovascular risk factors and the metabolic syndrome in pediatric nonalcoholic fatty liver disease. Circulation. 2008 Jul 15;118(3):277-83. doi: 10.1161/CIRCULATIONAHA.107.739920. Epub 2008 Jun 30. PMID 18591439
- [Background] Jin R, Le NA, Liu S, Farkas Epperson M, Ziegler TR, Welsh JA, Jones DP, McClain CJ, Vos MB. Children with NAFLD are more sensitive to the adverse metabolic effects of fructose beverages than children without NAFLD. J Clin Endocrinol Metab. 2012 Jul;97(7):E1088-98. doi: 10.1210/jc.2012-1370. Epub 2012 Apr 27. PMID 22544914
- [Background] Jin R, Welsh JA, Le NA, Holzberg J, Sharma P, Martin DR, Vos MB. Dietary fructose reduction improves markers of cardiovascular disease risk in Hispanic-American adolescents with NAFLD. Nutrients. 2014 Aug 8;6(8):3187-201. doi: 10.3390/nu6083187. PMID 25111123
- [Background] Schwimmer JB, Middleton MS, Behling C, Newton KP, Awai HI, Paiz MN, Lam J, Hooker JC, Hamilton G, Fontanesi J, Sirlin CB. Magnetic resonance imaging and liver histology as biomarkers of hepatic steatosis in children with nonalcoholic fatty liver disease. Hepatology. 2015 Jun;61(6):1887-95. doi: 10.1002/hep.27666. Epub 2015 Feb 5. PMID 25529941
- [Background] Jin R, Vos MB. Fructose and liver function--is this behind nonalcoholic liver disease? Curr Opin Clin Nutr Metab Care. 2015 Sep;18(5):490-5. doi: 10.1097/MCO.0000000000000203. PMID 26203597
- [Derived] Cohen CC, Li KW, Alazraki AL, Beysen C, Carrier CA, Cleeton RL, Dandan M, Figueroa J, Knight-Scott J, Knott CJ, Newton KP, Nyangau EM, Sirlin CB, Ugalde-Nicalo PA, Welsh JA, Hellerstein MK, Schwimmer JB, Vos MB. Dietary sugar restriction reduces hepatic de novo lipogenesis in adolescent boys with fatty liver disease. J Clin Invest. 2021 Dec 15;131(24):e150996. doi: 10.1172/JCI150996. PMID 34907907
- [Derived] Schwimmer JB, Ugalde-Nicalo P, Welsh JA, Angeles JE, Cordero M, Harlow KE, Alazraki A, Durelle J, Knight-Scott J, Newton KP, Cleeton R, Knott C, Konomi J, Middleton MS, Travers C, Sirlin CB, Hernandez A, Sekkarie A, McCracken C, Vos MB. Effect of a Low Free Sugar Diet vs Usual Diet on Nonalcoholic Fatty Liver Disease in Adolescent Boys: A Randomized Clinical Trial. JAMA. 2019 Jan 22;321(3):256-265. doi: 10.1001/jama.2018.20579. PMID 30667502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with NAFLD were recruited from two US academic clinical research centers (University of California, San Diego and Emory University)
Pre-assignment Details: Boys ages 11 - 16 with biopsy proven NAFLD were randomized
Groups:
- Intervention Group: Low free sugar diet
- Control Group: Habitual diet
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who consented to participate in the study and met eligibility criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.8 (1.8) | 13.4 (1.9) | 13.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 38
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 16 | 15 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Liver Fat Measured by Magnetic Resonance Imaging (MRI) in the Intervention Group Compared to Change in the Control Group
Description: The principal objective of this randomized and controlled pilot study is to evaluate whether 8 weeks of a low added sugar diet (<3%) in boys with NAFLD will change liver fat % measured by MRI.
Time Frame: Measurements done at baseline and week 8.
Measure: Mean (95% Confidence Interval); unit: Percentage of liver fat
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
Percentage of liver fat
  Baseline | 22.9 [18.7 to 28.0] | 19.4 [16.2 to 23.2]
  Week 8 | 14.9 [11.4 to 19.6] | 18.0 [14.0 to 22.4]

2. Secondary Outcome: Change in Alanine Aminotransferase (ALT) From Baseline to Week 8
Time Frame: Measurements done at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
U/L
  Baseline | 103.3 [79.7 to 133.8] | 81.8 [63.2 to 106.0]
  Week 8 | 61.3 [46.1 to 81.3] | 75.2 [56.7 to 99.9]

3. Secondary Outcome: Change in Aspartate Aminotransferase (AST) From Baseline to Week 8
Time Frame: Measurements doen at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
U/L
  Baseline | 52.0 [39.5 to 68.4] | 43.6 [33.2 to 57.4]
  Week 8 | 34.5 [27.3 to 43.6] | 39.1 [31.0 to 49.4]

4. Secondary Outcome: Change in Gamma-Glutamyl Transpeptidase (GGT) From Baseline to Week 8
Time Frame: Measurements done at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
U/L
  Baseline | 44.3 [33.5 to 58.6] | 44.1 [33.4 to 58.4]
  Week 8 | 33.0 [26.1 to 41.6] | 42.8 [33.9 to 54.0]

5. Secondary Outcome: Change in Insulin From Baseline to Week 8
Time Frame: Measurements done at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
mg/dL
  Baseline | 38.4 [28.6 to 51.6] | 41.8 [31.2 to 56.0]
  Week 8 | 37.7 [29.5 to 48.2] | 43.8 [34.5 to 55.5]

6. Secondary Outcome: Change in Homeostasis Model Assessment- Insulin Resistance (HOMA-IR) From Baseline to Week 8
Description: HOMA-IR was calculated as follows: fasting insulin (µU/mL) x fasting glucose (nmol/L)/22.5
Time Frame: Measurements done at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: HOMA score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
HOMA score
  Baseline | 8.6 [6.3 to 11.9] | 9.2 [6.7 to 12.7]
  Week 8 | 7.7 [5.9 to 10.0] | 10.2 [7.9 to 13.1]

7. Secondary Outcome: Change in Triglycerides From Baseline to Week 8
Time Frame: Measurements done at baseline and week 8
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
mg/dL
  Baseline | 121.7 [96.7 to 153.2] | 138.9 [110.3 to 174.8]
  Week 8 | 104.1 [82.6 to 131.3] | 134.3 [106.5 to 169.4]

ADVERSE EVENTS:
Time Frame: Adverse event details were collected throughout the duration of study participation, from the Baseline visit through the Week 8 follow up visit.
Description: For this study, an adverse event is considered any untoward medical occurrence in a subject participating in a clinical study that does not necessarily have a causal relationship with the dietary intervention.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=20) | Control Group (N=20)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Persistant Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02513121/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02513121/SAP_001.pdf